CLINICAL TRIAL: NCT01473186
Title: Prevalence of Menstrual Irregularities and Endometrial Pathology in Women Who Are Candidates for Bariatric Surgery: Correlation With Perceived Risk, Biomarkers, and Weight Loss
Brief Title: Study of Menstrual Irregularities and Endometrial Pathology in Women Undergoing Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Susan Modesitt, MD, Attending, University of Virginia
Other Study IDs: 15116
Record Dates: First submitted 2011-11-14; First posted 2011-11-17 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Morbid Obesity; Endometrial Pathology; Menstrual Irregularities
Keywords: morbid obesity; endometrial pathology; menstrual irregularities
MeSH Terms: conditions — Obesity, Morbid; Menstruation Disturbances

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, omentum, endometrium, adipose tissue
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Objectives: Given the profound impact of obesity on the genesis of endometrial cancer, this study proposes to prospectively evaluate the baseline prevalence of menstrual irregularities and endometrial pathology in morbidly obese women and discover risk stratification markers that can potentially identify the highest risk women who might benefit from targeted cancer prevention strategies in a future clinical trial.

* Specific Aim 1: To assess the prevalence of menstrual irregularities and to correlate gynecologic and menstrual history with the perceived personal risk and severity of gynecologic cancers in a population of female bariatric surgery candidates.
* Specific Aim 2: To determine the prevalence of endometrial hyperplasia and cancer in morbidly obese women undergoing bariatric surgery.
* Specific Aim 3: To obtain adipose, endometrium, and blood samples (before and after) bariatric surgery to assess baseline hormone levels and adipocyte-derived factors and to correlate with presence of menstrual irregularities, endometrial hyperplasia or cancer, and with postsurgical weight changes.

Methods:

* Specific Aim 1: After informed consent is obtained, a survey and medical history of prospective bariatric surgery patients will be performed at the University of Virginia.
* Specific Aim 2: For those women who undergo bariatric surgery, study investigators will perform endometrial biopsies at the time of bariatric surgery on participants to determine the status of the endometrial lining and the potential presence of endometrial cancer and its precursors.
* Specific Aim 3: At the time of surgery, blood, adipose, and endometrial tissue samples will collected for evaluation of adipocyte-related factors and correlation with clinical endpoints. Blood will also be collected at 6 and 12 months after surgery.

Anticipated results: This study will identify the prevalence and correlation of menstrual irregularities with endometrial abnormalities and cancer in morbidly obese women as well as define their perceived risk of developing cancer. Serum biomarkers in obese women with and without endometrial cancer/precancer would be evaluated for correlation and potential applicability for endometrial cancer screening in this high-risk population. Most importantly, this study may provide evidence as to whether screening (via endometrial biopsy or other serum markers) is warranted in asymptomatic, morbidly obese women and suggest potential preventive and risk reduction mechanisms.

DETAILED DESCRIPTION:
Obesity is defined qualitatively by the World Health Organization, is "abnormal or excessive fat accumulation that may impair health. Obesity is now estimated to lead to 280,000 deaths each year in the U.S., making it the second most common cause of preventable death only behind tobacco[1]. Obesity leads to an increased risk of several cancers, most notably endometrial cancer which is the fourth most common U.S. cancer with 40,000 affected women accounting for 6% of all estimated cancers in 2008 [2]. The recent increase in endometrial cancer has paralleled the increase in obesity [3]. The relative risk for an obese woman to develop endometrial cancer increases proportionally with increasing body mass index (BMI - weight in kilograms divided by height in meters squared)[4]. The risk may be 2-3 times [12,13] or up to 10-times greater for a woman more than 50 pounds overweight [5]. The most recent cohort study from Norway demonstrated increased adjusted relative risk based on BMI of 4.28 for a BMI of 35-39 and 6.36 for a BMI of 40 or over [6]. Morbidly obese women are also 23 fold more likely to harbor a precancerous endometrial condition compared to normal weight women [7]

The link of obesity with endometrial cancer has been well-established for over 20 years[5, 8]. For the most common histological subtype (endometrioid adenocarcinoma), the development of endometrial cancer is stimulated by the presence of estrogen. In obese patients, adipose tissue is responsible for elevating endogenous estrogen levels through its conversion of androgens to estrogens[9]. This also results in a relative decrease in progesterone, which normally 'protects' the uterine lining from over-stimulation by estrogen[8]. Obesity impacts multiple other factors including adiponectin, leptin, insulin, insulin growth factor one (IGF-1), tumor necrosis factor alpha (TNF-α), aromatase, and peroxisome proliferator activated receptor γ (PPAR) and the potential link of these factors to carcinogenesis has yet to be elucidated.

Propelled by increasing obesity, there is interest in identifying at risk populations who might benefit from screening and/or prevention. Viola et al looked at the prevalence of endometrial cancer and its precursors by biopsying 193 asymptomatic pre- and post-menopausal obese women (average BMI of 35.5 and 37.6 respectively) and found the prevalence of endometrial hyperplasia and cancer was 5.8% and 1% in premenopausal women and 12.1% and 3% in postmenopausal women[10]. These rates may even be higher in symptomatic women. For example, Schmeler et al evaluated 188 women diagnosed with endometrial cancer before age 50, 61% of the obese women had reported irregular menses, 14% a history of infertility, and 35% had diabetes[11]. The advantage to diagnosing endometrial cancer as precursor lesion or an early stage is due to a dramatic survival benefit; women with stage 1 disease have an excellent 5 year survival rate ranging between 80-95% and survival drops dramatically as stage increases. Women with earlier-stage disease generally need less-invasive and less-morbid post-operative treatments.

Universal screening of all women for endometrial cancer is not currently recommended[12, 13]. However, with the trend of endometrial cancer being found in younger, obese women, there is an increased likelihood that screening could decrease morbidity and mortality and that preventative strategies could be implemented in the highest risk women. Kwon and Lu conducted a cost-effectiveness analysis comparing no screening (standard of care), oral contraceptive pills as prevention, and endometrial biopsy either yearly or every other year after age 30. They concluded that the risk of endometrial cancer in a high risk population needed to be 13 times that of the general population to even warrant the use of oral contraceptives as a preventive measure [13]. Another cost analysis study confirmed that endometrial cancer screening is not warranted in the general population but that in a high risk population, annual serum screening might be efficacious and cost effective [12]. To date, there are no serum screening markers available in endometrial cancer. Prior authors have demonstrated that low adiponectin levels correlate with an increased rate of endometrial cancer. Adiponectin activates the AMPK pathway and the PPAR alpha pathway through two different receptors and functions to increase insulin sensitivity and decrease inflammation. Further prospective evaluation of adiponectin and other potential biomarkers is warranted in this population and to correlate with both obesity and weight loss[14-21].

Given that the prevalence of obesity continues to increase while the age at time of diagnosis of endometrial cancer has also begun to decrease, the early identification of cancer or pre-cancerous change of the uterus will become an important way to decrease morbidity and mortality in this ever-growing population of obese women[22, 23]. A previous retrospective study of women undergoing bariatric surgery at UVA demonstrated that endometrial cancer was one of the most common cancers diagnosed in this morbidly obese population, and that most women were diagnosed before their bariatric surgery at an average age of 35 and had a BMI of 65 kg/m2 [24]. Yet currently, the pre-operative gynecologic evaluation for bariatric surgery for weight loss includes only mammogram (to screen for breast cancer) and Pap smear (for cervical cancer) and compliance with these recommendations has not been well documented.

Given the profound impact of obesity on the genesis of endometrial cancer, this study proposes to prospectively evaluate the baseline prevalence of menstrual irregularities and endometrial pathology in morbidly obese women presenting for evaluation for bariatric weight loss surgery. The bariatric surgery population is ideal to define baseline characteristics of this population, to assess prevalence of endometrial abnormalities and to determine differences in hormones and adipocyte derived markers in women with and without endometrial abnormalities and to assess the impact of weight loss on these same markers. Ultimately, this study may allow the identification risk stratification markers that can potentially identify women who might benefit from targeted cancer prevention strategies in a future clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* female gender

Exclusion Criteria:

* male gender

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women who are candidates for bariatric surgery at the University of Virginia Center of Digestive health who are 18 or older
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Modesitt, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States